CLINICAL TRIAL: NCT01742143
Title: A Randomized Controlled Trial of the Impact of ICCAN on Cancer Treatment Completion and Quality of Life
Brief Title: Impact of ICCAN on Cancer Treatment Completion and Quality of Life
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The City College of New York (Other); Ralph Lauren Center for Cancer Care and Prevention (Other); Lincoln Medical and Mental Health Center (Other); Lutheran Medical Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: 12-223
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Cancer Patients
Keywords: Quality of life; cancer; 12-223
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Phase I: Refinement: 10 Black, Hispanic, and/or low-SES patients with TNBC (5 Spanish-speaking), will be recruited from MSK
  Interventions: Behavioral: The Integrated Cancer Care Access Network (ICCAN)
- Phase II, Arm 1: Usual and Customary Care (U&C): Participants in this group will receive the same referrals on social and economic resources as ICCAN group.
  Interventions: Behavioral: Usual and Customary Group (U&C)
- Phase II, Arm 2: ICCAN-IO: Arm 2 will consist of everything in Arm 1
  Interventions: Behavioral: The Integrated Cancer Care Access Network (ICCAN)

INTERVENTIONS:
Behavioral: The Integrated Cancer Care Access Network (ICCAN) — Patients will receive written materials on social and economic resources and services. Treatment Outcomes Survey at Intake, 3 mo, 6 mo, and 1 year.
  Chart review at 3 mo, 6 mo and 1 year, and as needed. Plus Initial needs assessment. Assistance with high priority social and economic needs.Monthly follow-up with ICCAN Access Facilitator to address ongoing needs in addition to as-needed assistance.
  Groups: Phase I: Refinement; Phase II, Arm 2: ICCAN-IO
Behavioral: Usual and Customary Group (U&C) — Patients will receive written materials on social and economic resources and services. Treatment Outcomes Survey at Intake, 3 mo, 6 mo, and 1 year.
  Chart review at 3 mo, 6 mo and 1 year, and as needed.
  Groups: Phase II, Arm 1: Usual and Customary Care (U&C)

SUMMARY:
The purpose of this 1 year study is to see if the ICCAN program is working, and to compare the ICCAN program to the standard hospital services provided in New York City hospitals, like meeting with a Social Worker or a Patient Navigator (a person who provides personal hospital guidance).

ELIGIBILITY:
Participant Inclusion Criteria:

Patient is eligible if he/she is

* fluent in English, Spanish, or Mandarin
* between the ages of 21-80 years old
* cancer patients currently receiving chemotherapy (started within the past month) and/or radiation therapy (started within the past week), or
* scheduled to begin chemotherapy and/or radiation therapy within the next 2 months (excluding surgery only patients)
* planning on remaining in the area for at least 1 year

Clinician is eligible if he/she:

* Has an MD or DO degree
* Is the treating physician providing care to a patient enrolled to the study

ICCAN-IO Phase 1: Refinement, participant is eligible if he/she per EMR or self-report:

* Is 18 - 85 years of age
* Has unresectable locally advanced, locally recurrent unresectable, metastatic, or high risk/early stage TNBC or stage I-IV lung cancer
* Eligible for FDA approved immunotherapy in the NYC metropolitan area (per self-report or per MSK patient EMR records).
* Is treated in the NY metropolitan area
* Self-identifies as Black or Hispanic, and/or is low-SES (low SES will be defined as household income < 200% of federal poverty level)
* Has English or Spanish proficiency
* Agrees to be audio-recorded

ICCAN-IO Phase 2: Pilot RCT, participant is eligible if he/she per EMR or self-report:

* Is 18 - 85 years of age
* Has stage II-III TNBC
* Treated at MSK Manhattan or OneMSK regional sites
* Self identifies as Black or Hispanic, and/or is low SES (low SES will be defined as household income < 200% of federal poverty level)
* Has English or Spanish proficiency
* Agrees to be audio-recorded

ICCAN-IO process evaluation study team participants only:

* Staff member who serves as an Access Facilitator
* Agrees to be audio-recorded

Participant Exclusion Criteria:

Patient is ineligible is he/she is:

* Presence of untreated psychiatric disturbance (i.e. acute psychiatric symptoms which require individual treatment) and/or cognitive impairment disorder (e.g., delirium or dementia) verified by medical record sufficient to preclude completion of the assessment measures, interview or informed consent

ICCAN-IO Phase 1: Refinement, participant is ineligible if he/she per EMR or self-report:

* Presence of untreated psychiatric disturbance (e.g., acute psychiatric symptoms which require individual treatment) and/or cognitive impairment disorder (e.g., delirium or dementia) sufficient to preclude completion of the assessment measures, interview or informed consent
* Participants or family members who are participating in MSK IHCD studies related to social determinants of health

ICCAN-IO Phase 2: Pilot RCT, participant is ineligible if he/she per EMR or self-report:

* Presence of untreated psychiatric disturbance (e.g, acute psychiatric symptoms which require individual treatment) and/or cognitive impairment disorder (e.g., delirium or dementia) sufficient to preclude completion of the assessment measures, interview or informed consent
* Participants or family members who are participating in MSK IHCD studies related to social determinants of health

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible cancer patients will be recruited in person by multilingual ICCAN Clinical Research Coordinators for participation in the study at Ralph Lauren Center for Cancer Care and Prevention (RLCCP), Lincoln Hospital (LH) and Lutheran Medical Center (LMC). In the event that MSK staff is not present when an eligible patient is identified. Refinement and Pilot RCT participants will be recruited through MSK Manhattan and OneMSK regional sites's.
Sampling Method: Probability Sample
Enrollment: 347 (Estimated)
Dates: Start 2012-11; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Treatment completion/adherence | 1 year
  The primary outcome, cancer treatment completion, will be determined by chart review at 3, 6, and 12 months after enrollment.

SECONDARY OUTCOMES:
Quality of life | 1 year
  depression, and stress (measured through validated scales included in the Cancer Treatment Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gany, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Lutheran Medical Center, Brooklyn, New York
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - City College of New York (Data Collection AND Data Analysis), New York, New York
  - Memorial Sloan Kettering at Ralph Lauren Center (Limited Protocol Activities), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York
  - Lincoln Hospital and Mental Health Center, The Bronx, New York

REFERENCES:
- [Derived] Gany F, Melnic I, Li Y, Finik J, Wu M, Ramirez J, Hwang C, Leng J, Blinder V. A Randomized Controlled Trial of the Integrated Cancer Care Access Network on Cancer Treatment Completion and Quality of Life. J Natl Compr Canc Netw. 2025 Jun 10;23(7):e257017. doi: 10.6004/jnccn.2025.7017. PMID 40494401
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/